CLINICAL TRIAL: NCT00203307
Title: A Single-Site, Double-Blind, Placebo-Controlled Cross-Over Trial Examining the Safety and Efficacy of Olanzapine Taken Daily for the Prevention of Episodic Migraine.
Brief Title: A Research Study Examining the Use of Olanzapine for the Prevention of Migraine
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Study terminated by sponsor
Sponsor: Thomas Jefferson University (Other)
Collaborators: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SDS/ZYP/02; 080-19000-H55901
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Results first posted 2011-08-10 (Estimated); Last update posted 2011-08-25 (Estimated); Status verified 2011-08

CONDITIONS: Migraine
MeSH Terms: conditions — Migraine Disorders

ARMS (2):
- Olanzapine then Placebo (Other): Olazepam
  Interventions: Drug: Olanzapine during first intervention period and placebo during second intervention period
- Placebo then olanzapine (Other)
  Interventions: Drug: Placebo during first intervention period, then olanzapine during second intervention period

INTERVENTIONS:
Drug: Olanzapine during first intervention period and placebo during second intervention period — Olanzapine (5-10 mg) daily during first intervention period, then placebo(matching)druing second intervention period (after a washout period)
  Arms: Olanzapine then Placebo
Drug: Placebo during first intervention period, then olanzapine during second intervention period — Placebo (matching) during first intervention period, then olanzapine (5-10 mg. daily) during the second intervention period (after a washout phase).
  Arms: Placebo then olanzapine

SUMMARY:
Olanzapine (o-lan-zah-peen) is a medication that has been approved by the Food and Drug Administration (FDA) for the treatment of patients with schizophrenia and/ or bipolar disorder. The trade name for this drug is Zyprexa®. Olanzapine has not been approved by the FDA for the prevention of migraine and is experimental for the purposes of this research study.

The Jefferson Headache Center at Thomas Jefferson University has developed this clinical study to evaluate the safety and effectiveness of Olanzapine in preventing migraine headaches.

ELIGIBILITY:
Inclusion Criteria:

* Subjects who are male or female between the ages of 18 and 65, inclusive
* Subjects who have a history of migraine with or without aura as defined by IHS criteria, for at least one year prior to screening
* Subjects who experience between 3 and 10 migraine attacks per month, for the three months preceding screening
* Subjects who have no more than 15 headache days per month
* Subjects who have been on a stable dose (no clinically significant changes) of all daily medications, for any indication, from 28 days prior to screening through the duration of the trial.
* Women who are using, or agree to use for the duration of the study, a medically acceptable form of contraception (as determined by the investigator), if female of childbearing potential.
* Subjects who are able to understand and comply with all study requirements
* Subjects who provide written informed consent prior to any study procedures being performed.

Exclusion Criteria:

* Women who are pregnant or lactating
* Subjects with an abnormal ECG that, in the investigators opinion, would expose them to increased risk of adverse events or interfere with study drug and/or analysis of efficacy/tolerability (subjects with QTC interval greater than 450ms will be excluded)
* Subjects currently taking, or have taken within the thirty days prior to screening, any neuroleptics > 1 day per week (such as Geodon, Zyprexa, Compazine, Phenergan, Seroquel and other drugs in the same class)
* Subjects currently taking or have taken within 4-weeks prior to screening any medication for the prevention of migraine
* Subjects who have failed more than two adequate trials of migraine prophylaxis, as determined by investigator
* Subjects who experience significant orthostatic hypotension, as determined by the investigator
* Subjects who, in the investigators opinion, have a history or have evidence of a medical condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial
* Subjects who, in the investigators opinion, have a history or have evidence of a psychiatric condition that would expose them to an increased risk of a significant adverse event or would interfere with the assessments of efficacy and tolerability during this trial.
* Subjects who have participated in an investigational drug trial in the 30 days prior to the screening visit

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 3 (Actual)
Dates: Start 2004-05; Primary Completion 2006-03 (Actual); Study Completion 2006-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Stephen D Silberstein, Principal Investigator — Thomas Jefferson University
Locations (1):
- Jefferson Headache Center, Philadelphia, Pennsylvania, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Olanzapine First, Then Placeb: Olanzapine (5-10 mg daily) during first intervention period and matching placebo in second intervention period (after washout period)
- Placebo First, Then Olanzapine: Matching placebo during first intervention period, then olanzapine (5-10 mg. daily) during second intervention period (after washout period).
Period: First Intervention
Arm/Group | Olanzapine First, Then Placeb | Placebo First, Then Olanzapine
Started | 3 (Double-blind cross-over design. Study terminated early. Results not analyzed.) | 0
Completed | 1 | 0
Not Completed | 2 | 0
Not completed — Adverse Event | 2 | 0
Period: Second Intervention
Arm/Group | Olanzapine First, Then Placeb | Placebo First, Then Olanzapine
Started | 1 (2 subjects dropped out of the 1st intervention period, due to fatugue.) | 0
Completed | 1 | 0
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Olanzapine First, Then Placeb | Placebo First, Then Olanzapine | Total
Number analyzed (Participants) | 3 | 0 | 3
Age Categorical [Number; unit: participants]
  <=18 years | 0 |  | 0
  Between 18 and 65 years | 3 |  | 3
  >=65 years | 0 |  | 0
Age Continuous [Mean (Standard Deviation); unit: years] | 50 (3) |  | 50 (3)
Gender [Number; unit: participants]
  Female | 2 |  | 2
  Male | 1 |  | 1
Region of Enrollment [Number; unit: participants]
  United States | 3 |  | 3

OUTCOME MEASURES:

1. Primary Outcome: Difference in Migraine Headache Periods During the Active Treatment Period as Compared to the Placebo Treatment Period, Per Subject.
Description: Definition of migraine headache period: One migraine period is defined as a 24-hour period starting at the time of onset of the migraine headache, during which the migraine headache is present*.
  Definition of time frames: First treatment period: Day 1 to 84. Second treatment period: day 113-196. Washout phase is day 85-112.
Time Frame: 84 day period on placebo compared to 84 day period on olanzapine
Measure: Mean (Standard Deviation); unit: headache periods
Arm/Group | Olanzapine First, Then Placeb | Placebo First, Then Olanzapine
Number analyzed (Participants) | 3 | 0
headache periods | 0 (0) |

2. Secondary Outcome: Reduction of Migraine Attack Frequency During Each 28-day Interval of the Active Treatment Period as Compared to Each 28-day Interval of the Placebo Treatment Period, Per Subject. Individual Migraine Attacks Are Separated by 48-hours Pain Free Time. A
Time Frame: each 28 day interval of active treatment c ompared to placebo
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: migraine attacks

3. Secondary Outcome: Reduction in Days Using an Acute Headache Treatment During the Active Treatment Period as Compared to the Placebo Treatment Period, Per Subject.
Time Frame: 84 day period on olanzapine compared to 84 day period on placebo
Reporting Status: Not Posted
Measure: Mean (Standard Deviation); unit: days

ADVERSE EVENTS:
Arm/Group | Olanzapine First, Then Placeb | Placebo First, Then Olanzapine
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/0
Other Adverse Events (participants affected / at risk) | 2/3 | 0/0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Olanzapine First, Then Placeb (N=3) | Placebo First, Then Olanzapine (N=0)
lethargy (Nervous system disorders) | 2 | 0 (0) — 2 subjects withdrew from study before completion due to lethargy

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes